CLINICAL TRIAL: NCT00072228
Title: Phase I Study of Soblidotin and Gemcitabine in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Soblidotin and Gemcitabine in Treating Patients With Locally Advanced or Metastatic Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: DAIICHI-1027A-PRT008; CDR0000339345 (Registry Identifier: PDQ (Physician Data Query)); CPMC-IRB-20031085; NCT00072228
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2006-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Gemcitabine; soblidotin; Drug Therapy

INTERVENTIONS:
Drug: gemcitabine
Drug: soblidotin
Procedure: chemotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as soblidotin and gemcitabine, use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of soblidotin and gemcitabine in treating patients with locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of soblidotin and gemcitabine in patients with locally advanced or metastatic solid tumors.
* Determine the dose-limiting toxic effects of this regimen in these patients.

Secondary

* Determine the toxicity profile of this regimen in these patients.
* Determine the pharmacokinetics of this regimen in these patients.
* Determine, preliminarily, the antitumor activity of this regimen in these patients.

OUTLINE: This is an open-label, nonrandomized, multicenter, dose-escalation study.

Patients receive gemcitabine IV over 30 minutes and soblidotin IV over 1 hour on days 1 and 8. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of soblidotin and gemcitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed for survival every 3 months after completion of study therapy.

PROJECTED ACCRUAL: Approximately 35 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed locally advanced or metastatic solid tumors
* Minimally pretreated
* Not refractory to prior gemcitabine therapy
* No disease progression during initial treatment with gemcitabine
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT or SGPT no greater than 2.5 times ULN (5 times ULN if liver metastases are present)

Renal

* Creatinine no greater than 1.5 times ULN

Cardiovascular

* Ejection fraction at least 40% by MUGA

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No psychiatric disorder that would preclude study consent or compliance
* No concurrent severe or uncontrolled underlying medical disease unrelated to the tumor that would compromise patient safety or affect study outcome
* No hypersensitivity to gemcitabine
* No other malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix unless in complete remission and off all therapy for that disease for at least 2 years
* No serious infection
* No grade 2 or greater neuropathy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent anticancer biologic therapy

Chemotherapy

* See Disease Characteristics
* Recovered from prior chemotherapy
* No other concurrent anticancer chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Recovered from prior radiotherapy
* No concurrent anticancer radiotherapy
* Concurrent localized palliative radiotherapy to a non-indicator lesion for pain control allowed only if other methods of pain control are ineffective

Surgery

* At least 4 weeks since prior major surgery and recovered

Other

* More than 28 days since prior investigational drugs, including analgesics or antiemetics
* At least 4 weeks since prior myelosuppressive therapy
* No other concurrent anticancer therapy
* No other concurrent anticancer cytotoxic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. DeJager, MD, FACP, Study Chair — Daiichi Pharmaceuticals
Locations (2):
- United States (2):
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York